CLINICAL TRIAL: NCT00967109
Title: Establishment of Optimal Transfusion Threshold During Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Kamilla Nielsen, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H-C-2009-072
Record Dates: First submitted 2009-08-24; First posted 2009-08-27 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Anemia; Spine Surgery
Keywords: Anemia; Tissue oxygenation; Spine surgery
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allowed drop in hemoglobin to 4,5-5,5 mmol/L (Active Comparator): Transfusion with red blood cells to level between 4.5-5.5 mmol/L
  Interventions: Other: Allowed drop in hemoglobin to level between 4,5-5,6 mmol/L
- Allowed drop in hemoglobin to 5,5-6,5 mmol/L (Experimental): Transfusion with red blood cells to level between 5.5-6.5 mmol/L
  Interventions: Other: Allowed drop in hemoglobin to level between 5,6-6,5 mmol/L

INTERVENTIONS:
Other: Allowed drop in hemoglobin to level between 4,5-5,6 mmol/L — Transfusion with red blood cells to hemoglobin level between 4,5-5,5 mmol/L
  Arms: Allowed drop in hemoglobin to 4,5-5,5 mmol/L
Other: Allowed drop in hemoglobin to level between 5,6-6,5 mmol/L — Transfusion with red blood cells to hemoglobin level between 5,6-6,5 mmol/L
  Arms: Allowed drop in hemoglobin to 5,5-6,5 mmol/L

SUMMARY:
The purpose of this study is to determine whether a higher threshold for transfusion with red blood cells improves the tissue oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients undergoing spine surgery
* Be legally competent
* Read and understand Danish

Exclusion Criteria:

* Present malignant disease
* Previously apoplexia cerebri
* Known heart disease with functionality equivalent to NYHA II or CCS II or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The change in subcutaneous oxygen tension from incision. | Every fifteen minutes throughout surgery
  The primary endpoint is the change in subcutaneous oxygen tension from incision until the time most patients is still undergoing surgery. Subcutaneous oxygen tension is measured every fifteen minutes throughout surgery. The oxygen tension is measured with a polygraphic electrode (Clark's electrode).

SECONDARY OUTCOMES:
Oxygenation of the brain | Every fifteen minutes throughout surgery
The concentration of lactate in plasma | Every half an hour throughout surgery
Variation in the ST-segment of the ECG | Every fifteen minutes throughout surgery
Muscular saturation of the deltoid muscle | Every fifteen minutes throughout surgery
  The change in muscular saturation from incision until the time when most patientes are still undergoing surgery. Furthermore the lowest measured and the last measured muscular saturation is also evaluated.
The change in subcutaneous oxygen tension from incision. | Every fifteen minutes throughout surgery
  The lowest measured subcutaneous oxygen tension and the last measured subcutaneous oxygen tension throughout surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla Nielsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark